CLINICAL TRIAL: NCT01699425
Title: Multicentric Comparative Randomized Study of the Single-incision Sling Ajust® Versus Suburethral Transobturator Slings.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Hospital Universitari de Bellvitge (Other); Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other); Hospital de Viladecans (Other); Serveis de Salut Integrats Baix Empordà (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AJA201205
Record Dates: First submitted 2012-09-22; First posted 2012-10-03 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Female Stress Urinary Incontinence
Keywords: Stress urinary incontinence.; Suburethral sling.; Single-incision suburethral sling.; Ajust.; Transobturator tape.
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Ajust (Experimental): Experimental group: surgery to treat stress urinary incontinence with the sling Ajust®
  Interventions: Device: Ajust sling
- Classical transobturator tape (Active Comparator): Control group: surgery to treat stress urinary incontinence with the Align® sling.
  Interventions: Device: Classical transobturator sling

INTERVENTIONS:
Device: Ajust sling
  Arms: Ajust
Device: Classical transobturator sling — Control group
  Other Names: Align®
  Arms: Classical transobturator tape

SUMMARY:
The transobturator tension-free vaginal tape (TOT) procedure has demonstrated high cure rates comparable to those obtained by retropubic suburethral tape, becoming the first line treatment for stress urinary incontinence (SUI) in many cases. The TOT procedure is not exempt from complications such as bleeding, bladder injuries and pain in the thigh/groin. In addition it is commonly performed under general or regional anesthesia1-3. The single-incision mini-slings (SIMS) were developed to reduce the risk of complications by avoiding the blind passage of the trocars through the obturator space. In addition, the use of SIMS could enable surgeons to perform the procedure truly under local anesthesia.

Different devices for SIMS procedure are available. However, the evidence about their efficacy is controversial4-7. The main limitation of these devices could be the predetermined length of the mesh and the weakness on its fixation. The design of the SIMS Ajust® allows adjusting the length of the sling to each individual woman and provides a robust fixation into the obturator membrane. Recent prospective studies on the efficacy and safety of the sling Ajust® have obtained promising results8,9. Even so, the NICE guidelines advise to use SIMS in the context of research studies10.

The objective of this study is to establish if the effectiveness of the SIMS Ajust® is non-inferior to that of a standard TOT, as well as to compare the comorbidity of both procedures. Owing to the new appearance and fast evolution of these procedures, randomized comparative studies with SIMS are required in order to determine its place in the treatment of SUI.

ELIGIBILITY:
Inclusion Criteria:

* Stress urinary incontinence with urethral hypermobility.

Exclusion Criteria:

* Incapacity to understand the information or give their consent.
* Previous anti-incontinence surgery with slings.
* Urethral hypomobility (Q-tip test <30º).
* Low pressure urethra (MUCP < 20cmH2O).
* Detrusor overactivity.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Comparison of the cure rates between the single incision sling Ajust and classical transobturator tapes. | Up to one year
  Percentage of patients who are regarded as cured or improved based on the following criteria:
  * Improvement on the International consultation on Incontinence Urinary Questionnaire-Short Form 1 year after the surgery.
  * Negative Cough Stress test 1 year after surgery.

SECONDARY OUTCOMES:
Number of participants with adverse events | 0, 1, 6 and 12 months after surgery
  Comparison of the intra- and postoperative complications between procedures

OTHER OUTCOMES:
Change in the Maximal Urethral Closure Pressure. | One year after surgery.
  Comparison of the changes in the Maximal Urethral Closure Pressure (cmH2O) measured preoperatively and 1 year after surgery.

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Hospitalet, Barcelona
  - Hospital de Viladecans, Viladecans, Barcelona
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona, Girona
  - Hospital de Palamós, Palamós, Girona